CLINICAL TRIAL: NCT05710731
Title: The Effects of Virtual Reality Simulation, Computer Based Simulation and Low Reality Simulation Methods Used in Urinary Catheterization Training on Skills, Satisfaction and Self-Confidence in Nursing Students
Brief Title: The Urinary Catheterization Training on Skills, Satisfaction and Self-Confidence in Nursing Students
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cukurova University (Other)
Collaborators: The Scientific and Technological Research Council of Turkey (Other)
Responsible Party: Principal Investigator, ECE KURT, lecturer, Cukurova University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: Cukurova Ece Kurt SBF 01
Record Dates: First submitted 2023-01-14; First posted 2023-02-02 (Actual); Last update posted 2023-02-02 (Actual); Status verified 2023-01

CONDITIONS: Catheter-Related Infections; Urinary Catheterization
MeSH Terms: conditions — Catheter-Related Infections

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- low-reality simulation Group (Experimental): In this group, urinary catheterization will be performed through a plastic half-hip model.
  Interventions: Other: Use of simulation in urinary catheterization training
- Computer Based Simulation Group (Experimental): In this group, urinary catheterization will be performed through a computer-based full-body model.
  Interventions: Other: Use of simulation in urinary catheterization training
- Virtual Reality Simulation Group (Experimental): In this group, urinary catheterization will be performed through a software based on virtual reality technology.
  Interventions: Other: Use of simulation in urinary catheterization training

INTERVENTIONS:
Other: Use of simulation in urinary catheterization training — To train students on urinary catheterization by using one of 3 different simulation methods.

SUMMARY:
In our study, it is planned to use three different simulation methods. One of these; It is a low-reality simulator, a hip model. It is known that this model is used by many universities in nursing education today and is called the traditional method. Both of the other simulators the investigators will use are high-fidelity models. One of them is a computer-based full-body manikin and the other is a virtual reality simulation.

DETAILED DESCRIPTION:
The research was designed as a randomized controlled experimental study to determine the effects of virtual reality simulation, computer-based simulation and low-reality simulation methods used in urinary catheterization training on skills, satisfaction and self-confidence in nursing students. The research will be carried out in Çukurova University Health Sciences Faculty Nursing Department Vocational Skills Laboratory in the spring semester of 2022-2023 academic year. The students who will participate in the research do not have clinical practice experience yet.

The computer-based simulation model (S550.100 Noelle, Gynecology Model) to be used in our study consists of the full human body and can produce real human sounds (pain response, fear, etc.). Thus, thanks to the computer connection, the communication between the student and the simulator is increased and the reality of the clinical environment is maintained. Person performing urinary catheterization on the simulator; can feel the resistance of structures such as urethra, sphincter and bladder, which are similar to the anatomical structure of the real patient. When the catheter enters the bladder, as in a real patient, artificial urine (yellow water) flows through the catheter and the catheter balloon can be fully inflated/deflated during catheter insertion/removal.

Considering the technical features of the virtual reality simulator, which is another simulator to be used in our study; Thanks to the glasses used, it is possible to say that the patient and hospital environment are presented to the students in 3D with high reality. With the use of glasses, students will be able to perform urinary catheterization with the joysticks they hold in their hands. Thanks to this technology, it is possible for students to evaluate themselves by facing situations that are difficult to control in real life, as if they are actually experiencing them, to gain the right knowledge and skills through the mistakes they have made, and to gain experience by developing their sense of confidence.

Another simulator to be used in the study is a low-reality hip model. This is a model used to gain the ability to apply urinary catheterization and only female external reproductive organs can be seen. While the catheter moves through the urinary system and enters the bladder, the feeling of resistance and pressure experienced on real patients cannot be experienced. After the catheter is integrated into the external reproductive organ, operations such as seeing its progress along the urethra and bladder, controlling its location and inflating the balloon cannot be performed. It is the traditional method used for urinary catheterization practice training of nursing students.

The sample size was calculated by Power analysis (G*Power 3.1.9.2) based on a similar study done before. Based on the results of students' self-confidence and satisfaction levels, a total of 156 samples were determined for each group with a test power of 0.80, 95% confidence (1-α) and an effect size of f=0.25, with a minimum of 53 samples. identified as a student. In the 2022-2023 academic year, the Department of Nursing enrolled 182 students in the first class. All students who meet the criteria to participate in the research will be assigned to one of the three simulation groups using simple random sampling method. Students will be listed taking into account the last three digits of the school number. The web address https://www.randomizer.org will be used for random assignment.

ELIGIBILITY:
Inclusion Criteria:

* To register for the Nursing Fundamentals II Course for the first time,
* Volunteering to participate in the research,

Exclusion criteria from the study:

* To be a graduate of Health Vocational High School,
* Working as a nurse/midwife
* Have any previous experience of urinary catheterization,

Exclusion Criteria:

* Not attending the theoretical lesson,
* Not participating in demonstration and group work,
* Not participating in skill measurements

Ages: 18 Years to 24 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 156 (Estimated)
Dates: Start 2023-02-14 (Estimated); Primary Completion 2023-02-28 (Estimated); Study Completion 2023-04-04 (Estimated)

PRIMARY OUTCOMES:
Urinary Catheterization Practice Skills Evaluation | 10 minutes
  -Each student's urinary catheterization practice will be video-recorded one by one by the researcher, and then the videos will be watched and the "Urinary Catheterization Skills Checklist" will be filled.

SECONDARY OUTCOMES:
Student Satisfaction and Self Confidence Measurement | 10 minutes
  - At the end of the application, students will fill in the "Student Satisfaction and Self Confidence in Learning Scale".

OTHER OUTCOMES:
Simulation Design Evaluation | 10 minutes
  At the end of the application, students will fill in the "Simulation Design Scale".

IPD SHARING:
Plan to Share IPD: No